CLINICAL TRIAL: NCT07323277
Title: The Effect of Smoking on Macrophage Polarization in the Pathogenesis of Periodontitis
Brief Title: Effect of Smoking on Macrophage Polarization in Periodontitis
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Asli Ege Ozdamar, PhD Candidate / Principal Investigator, Suleyman Demirel University
Other Study IDs: SDU-Perio-iNOS-ARG1-01; TDK-2024-9512 (Other: SDU BAP)
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis
Keywords: Smoking; Macrophage Polarization; M1/M2 Macrophages; iNOS; Arginase-1; Periodontal Inflammation; Periodontal Disease
MeSH Terms: conditions — Periodontitis; Smoking; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival tissue biopsies (approximately 2×2 mm) collected during periodontal surgical procedures performed after completion of Phase I periodontal therapy. Samples were immediately stored at -80 °C and used for ELISA analysis of iNOS and Arginase-1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Non-Smokers: Systemically healthy individuals who do not smoke and present with clinically healthy periodontal status. Gingival tissue samples were collected after completion of Phase I periodontal therapy during routine periodontal procedures.
- Periodontitis Non-Smokers: Systemically healthy individuals diagnosed with periodontitis who do not smoke. Gingival tissue biopsies were obtained after completion of Phase I periodontal therapy during periodontal surgical procedures.
- Healthy Smokers: Systemically healthy individuals who smoke (≥10 cigarettes/day) and exhibit clinically healthy periodontal status. Gingival tissue samples were collected after completion of Phase I periodontal therapy during periodontal procedures.
  Interventions: Other: Smoking Exposure
- Periodontitis Smokers: Systemically healthy individuals who smoke (≥10 cigarettes/day) and are clinically diagnosed with periodontitis. Gingival tissue samples were collected after completion of Phase I periodontal therapy during periodontal surgical procedures.
  Interventions: Other: Smoking Exposure

INTERVENTIONS:
Other: Smoking Exposure — Exposure to cigarette smoking, defined as smoking ≥10 cigarettes per day. Participants were classified as smokers or non-smokers based on self-reported smoking status.
  Groups: Healthy Smokers; Periodontitis Smokers

SUMMARY:
This observational case-control study investigates the effect of smoking on macrophage polarization in the pathogenesis of periodontitis. Adult participants who were either systemically healthy smokers or non-smokers, and who met the clinical criteria for periodontal health or periodontitis, were included. Gingival tissue samples were collected during periodontal procedures performed after completion of Phase I periodontal therapy, and the expression levels of macrophage polarization markers (iNOS and Arginase-1) were analyzed using ELISA. In addition, comprehensive clinical periodontal measurements-including probing pocket depth, clinical attachment level, bleeding on probing, Plaque Index, and Gingival Index-were recorded to evaluate the relationship between smoking status, inflammatory burden, and macrophage phenotype. The study aims to clarify how smoking modulates the balance between M1 and M2 macrophage responses in periodontal tissues.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease in which macrophage polarization plays a key regulatory role in the host immune response. Smoking is a well-established risk factor that alters inflammatory pathways and immune cell behavior. This study was designed to examine how smoking influences macrophage polarization-specifically the balance between M1 (iNOS-mediated) and M2 (Arginase-1-mediated) phenotypes-in periodontal tissues.

Systemically healthy adult participants were recruited and categorized into four groups based on smoking status and periodontal condition: (1) healthy non-smokers, (2) periodontitis non-smokers, (3) healthy smokers, and (4) periodontitis smokers. Gingival tissue samples (approximately 2×2 mm) were collected during periodontal surgical procedures performed after completion of Phase I periodontal therapy, immediately stored at -80 °C, and processed for biochemical analysis. Comprehensive clinical periodontal measurements-including probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), Plaque Index (PI), and Gingival Index (GI)-were recorded on the same day to evaluate periodontal status and inflammatory burden. ELISA was used to quantify iNOS and Arginase-1 levels in gingival tissues.

The primary objective of this study is to determine whether smoking shifts the macrophage phenotype toward a more pro-inflammatory M1 profile or suppresses M2-associated regulatory pathways in the context of periodontitis. The findings are expected to contribute to a better understanding of smoking-related alterations in periodontal immune mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of volunteer participants aged 18-65 years who were referred to the Department of Periodontology at Süleyman Demirel University Faculty of Dentistry for periodontal treatment and who met the inclusion criteria without violating any exclusion criteria.

Exclusion Criteria:

* Individuals who did not consent to participate in the study
* History of any periodontal treatment within the past 6 months
* Use of systemic antibiotics within the past 3 months
* Pregnancy or lactation
* Psychological or physical conditions that may interfere with cooperation during clinical examination
* History of substance or alcohol abuse
* Presence of severe malocclusion or ongoing orthodontic treatment
* Acute dental pain due to caries, abscess, or other odontogenic infections
* Presence of systemic diseases with oral manifestations or any systemic condition known to affect periodontal tissues
* History of malignancy
* Use of medications that can influence periodontal parameters (e.g., anti-inflammatory drugs) within the past 3 months
* Participation in another scientific or clinical research study within the past 3 months

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of systemically healthy volunteer adults aged 18-65 years who presented to the Periodontology Clinic of Süleyman Demirel University Faculty of Dentistry with a need for periodontal treatment. Eligible participants were assigned to one of four groups based on smoking status and periodontal condition: healthy non-smokers, periodontitis non-smokers, healthy smokers, and periodontitis smokers. All participants were evaluated according to the study's predefined inclusion and exclusion criteria before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Gingival iNOS Level | At the time of periodontal surgery following completion of Phase I periodontal therapy.
  Concentration of inducible nitric oxide synthase (iNOS) in gingival tissue biopsies measured by ELISA (ng/mg tissue).
Gingival Arginase-1 Level | At the time of periodontal surgery following completion of Phase I periodontal therapy.
  Concentration of Arginase-1 in gingival tissue biopsies measured by ELISA (ng/mg tissue).

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) | Immediately prior to periodontal surgery, following completion of Phase I periodontal therapy.
  Mean probing pocket depth (mm) recorded at six sites per tooth using a periodontal probe.
Clinical Attachment Level (CAL) | Immediately prior to periodontal surgery, following completion of Phase I periodontal therapy.
  Clinical attachment level (mm) recorded at six sites per tooth using a periodontal probe.
Bleeding on Probing (BOP) | Immediately prior to periodontal surgery, following completion of Phase I periodontal therapy.
  Bleeding on probing percentage calculated as the proportion of bleeding sites to total sites examined.
Plaque Index (PI) | Immediately prior to periodontal surgery, following completion of Phase I periodontal therapy.
  Dental plaque accumulation assessed using the Silness and Löe Plaque Index. Plaque scores were recorded at four surfaces per tooth and scored on a scale from 0 to 3, where 0 indicates no plaque and 3 indicates abundant plaque accumulation. Higher scores indicate worse plaque status.
Gingival Index (GI) | Immediately prior to periodontal surgery, following completion of Phase I periodontal therapy.
  Gingival inflammation assessed using the Löe and Silness Gingival Index. Gingival Index scores were recorded at four surfaces per tooth and scored on a scale from 0 to 3, where 0 indicates normal gingiva and 3 indicates severe gingival inflammation. Higher scores indicate worse gingival status.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal YETKİN AY, Prof. Dr., Principal Investigator — Süleyman Demirel University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Süleyman Demirel University Faculty of Dentistry, Department of Periodontology, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study is a single-center thesis research project, and data sharing is not permitted under institutional and ethical regulations.